CLINICAL TRIAL: NCT01743937
Title: A Randomized, Controlled, Open Label Trial Comparing the Ischemic Preconditioning Effects of Ticagrelor and Clopidogrel in Humans
Brief Title: A Trial Comparing the Ischemic Preconditioning Effects of Ticagrelor and Clopidogrel in Humans
Acronym: ETCH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor terminated due to budgetary issue
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, James De Lemos, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZUTSW
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Ischemic Preconditioning
Keywords: Ischemic preconditioning; Ticagrelor; Antiplatelet therapy; Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Active Comparator): Coronary occlusion with balloon inflation
  Interventions: Procedure: Coronary occlusion with balloon inflation
- Clopidogrel (Active Comparator): Coronary occlusion with balloon inflation
  Interventions: Procedure: Coronary occlusion with balloon inflation

INTERVENTIONS:
Procedure: Coronary occlusion with balloon inflation

SUMMARY:
Antiplatelet therapy remains a cornerstone in the treatment of acute and chronic coronary artery disease. Aspirin was the first such therapy to prove its benefits in acute myocardial infarction. Compared to aspirin monotherapy, the combination of aspirin and clopidogrel, a thienopyridine P2Y12 inhibitor, has been demonstrated to reduce adverse event rates among patients with acute coronary syndromes (with or without ST-segment elevation) and those receiving intracoronary stents. In the Triton-TIMI 38 trial a novel thienopyridine, prasugrel, was compared to clopidogrel in patients with acute coronary syndrome undergoing percutaneous coronary intervention. Although prasugrel significantly reduced recurrent myocardial infarction, bleeding rates were increased and no improvement in cardiac or all-cause mortality was demonstrated. However, in 2009, the authors of the PLATO trial demonstrated an unexpected cardiovascular mortality benefit with ticagrelor over clopidogrel, an endpoint not previously met by any other antiplatelet agent against an active comparator. Based on the reproducible adverse events seen in the DISPERSE, DISPERSE-2, and PLATO trials, an adenosine-mediated effect of ticagrelor is proposed.

Hypothesis: The aim of this study is to test the hypothesis that ticagrelor produces pharmacologic ischemic preconditioning, an undescribed potential off-label property of ticagrelor that could represent a plausible mechanism for its effects on cardiovascular mortality.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing clinically-indicated PCI for stable or progressive exertional angina without rest angina, ST-segment shift, or elevated CK-MB or troponin-T or I
* Willing and able to give informed consent and to comply with study procedures
* Found to have single or two-vessel obstructive, non-occlusive (≥ 70% but < 100% stenosis), coronary artery disease with plans for treatment of all lesions by PCI
* Target lesion location in the proximal or mid coronary vessel with reference diameter ≥ 2.5 mm

Exclusion Criteria:

* Known allergy to aspirin, clopidogrel, or ticagrelor
* Need for concomitant cardiac procedure, such as valve repair or replacement
* Age ≥ 75
* Concomitant theophylline/aminophylline use
* Baseline ECG with infarct or conduction abnormalities (i.e. LVH with repolarization abnormality, bundle branch block, ST-segment abnormalities)
* Presenting with an ST-segment elevation or non ST-segment elevation myocardial infarction
* Evidence of prior myocardial infarction by cardiac imaging
* Depressed left ventricular systolic function (ejection fraction < 50%)
* Clinical congestive heart failure
* End-stage renal disease
* Presence of coronary collaterals on diagnostic coronary angiography
* Presence of coronary thrombus on diagnostic coronary angiography
* Diffuse obstructive disease (≥ 70% stenosis) in the distal segment of the target vessel
* Left main and/or three-vessel coronary artery disease
* Concomitant need for Warfarin therapy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Degree of ST-segment elevation by intracoronary ECG during coronary balloon inflation | 7-12 days after drug randomization

SECONDARY OUTCOMES:
Degree of ST-segment elevation by surface ECG during coronary balloon inflation | 7-12 days after drug randomization
Maximum inflation time tolerated following coronary balloon inflation | 7-12 days after drug randomization
  This is defined as the amount of time the patient tolerates having loss of coronary flow in the target coronary artery during balloon inflation.
Time to ST-segment elevation during coronary balloon inflation | 7-12 days after drug randomization
Angina score during coronary balloon inflation | 7-12 days after drug randomization
  This will be reported by the study subject during coronary balloon occlusion based on a validated pain scale.
Wall motion on chest wall echocardiography before and during coronary balloon inflation | 7-12 days after drug randomization
Strain rate on chest wall echocardiography before and during coronary balloon inflation | 7-12 days after drug randomization

CONTACTS AND LOCATIONS:
Overall Officials: James de Lemos, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Dallas Veterans Affairs Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas